CLINICAL TRIAL: NCT02973841
Title: Sono-ease Device for Internal Jaguar Vein Cannulation
Acronym: Sono-ease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, lecturer of anesthesia, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sono-ease
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Internal Jugular Vein Cannulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sono-ease group (Experimental): insertion IJV catheter using sono-ease device
  Interventions: Device: Sono-ease device

INTERVENTIONS:
Device: Sono-ease device — insertion of US guided IJV using sono-ease device

SUMMARY:
A novel device attached to ultrasound probe designed to increase success rate and safety of internal jugular vein cannulation.

ELIGIBILITY:
Inclusion Criteria:

* all patients indicated for IJV catheterization

Exclusion Criteria:

* neck deformities-coagulopathy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
complications rate | 24 hours
  hematoma-arterial puncture-pneumothorax

IPD SHARING:
Plan to Share IPD: Yes